CLINICAL TRIAL: NCT02811211
Title: A Noninterventional Genotype/Phenotype Study of mGluR Mutations in Children and Adolescents With Attention Deficit Hyperactivity Disorder (ADHD)
Brief Title: A Noninterventional Genotype/Phenotype Study of mGluR Mutations in Children and Adolescents With ADHD
Status: Completed | Type: Observational
Sponsor: Aevi Genomic Medicine, LLC, a Cerecor company (Industry)
Responsible Party: Sponsor
Organization: Avalo Therapeutics, Inc. (Industry)
Other Study IDs: MDGN-NFC1-ADHD-001
Record Dates: First submitted 2016-06-21; First posted 2016-06-23 (Estimated); Last update posted 2021-07-06 (Actual); Status verified 2017-02

CONDITIONS: Attention Deficit Disorder With Hyperactivity
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Saliva
Oversight: Data Monitoring Committee: No

SUMMARY:
This noninterventional study will assess genomic changes in the metabotropic glutamate receptor (mGluR) network in children and adolescents with ADHD.

DETAILED DESCRIPTION:
Male and female subjects 6 to 17 years of age with a primary psychiatric diagnosis of ADHD will be enrolled in this study. The subject and his or her parent/guardian must agree to genotyping to determine whether the subject has disruptive mutations within any of the approximately 274 mGluR-network genes, and complete an interview that will include information about the subject's ADHD history, treatment, and co-morbidities.

ELIGIBILITY:
Inclusion Criteria:

* The subject is male or female ≥6 and ≤17 years of age.
* The subject has ADHD as defined by the Diagnostic and Statistical Manual of Mental Disorders, 5th edition.
* The subject, his or her legally responsible representative, and investigator agree to complete ADHD history, treatment, and comorbidity electronic case report form (eCRF).

Exclusion Criteria:

* The subject or parent/legal guardian is in the opinion of the investigator mentally or legally incapacitated and unable to provide informed consent/assent for participation in the study.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Subjects between the ages of 6 years and 17 years of age with a previously established diagnosis of ADHD will be eligible for screening.
Sampling Method: Non-Probability Sample
Enrollment: 1894 (Actual)
Dates: Start 2016-02; Primary Completion 2017-01-06 (Actual); Study Completion 2017-01-06 (Actual)

PRIMARY OUTCOMES:
Presence of mGluR network mutations | At study enrollment

CONTACTS AND LOCATIONS:
Locations (1):
- A.I. DuPont Hospital for Children, Wilmington, Delaware, United States

IPD SHARING:
Plan to Share IPD: Undecided